CLINICAL TRIAL: NCT01622088
Title: An Open-Label, Multicenter, Extension Study to Evaluate the Long-Term Safety and Efficacy of Dexpramipexole (BIIB050) in Subjects With Amyotrophic Lateral Sclerosis
Brief Title: Phase 3 Extension Study of Dexpramipexole in ALS
Acronym: ENVISION
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The Initial Phase 3 Study (NCTO1281189) did not meet its primary efficacy endpoint.
Sponsor: Knopp Biosciences (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 223AS304; EUDRA CT #: 2011-006119-70
Record Dates: First submitted 2012-05-03; First posted 2012-06-18 (Estimated); Results first posted 2022-04-07 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS, Motor Neuron Disease, Amyotrophic Lateral Sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Dexpramipexole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dexpramipexole (Experimental): Dexpramipexole open-label
  Interventions: Drug: Dexpramipexole

INTERVENTIONS:
Drug: Dexpramipexole — Oral tablet 150 mg given twice daily (BID)
  Other Names: BIIB050

SUMMARY:
The purpose of the study is to collect long-term safety data from subjects with Amyotrophic Lateral Sclerosis (ALS) exposed to dexpramipexole.

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS) is a rapidly progressive, degenerative disease of motor neurons in the brain and spinal cord that leads to muscle atrophy and spasticity in limb and bulbar muscles resulting in weakness and loss of ambulation, oropharyngeal dysfunction, weight loss, and ultimately respiratory failure. The purpose of this study is to collect long-term safety data from subjects with Amyotrophic Lateral Sclerosis (ALS) exposed to dexpramipexole.

ELIGIBILITY:
Inclusion Criteria:

* Subject has the ability to understand the purpose and risks of the study and provide signed and dated informed consent (or have the consent confirmed by a witness if unable to write) and authorization to use protected health information (PHI) in accordance with national and local subject privacy regulations.
* Subject was enrolled in either CL211 (NCT00931944) or Study 223AS302 (NCTO1281189).
* Subject has completed their last visit in Study CL211 (NCT00931944) or Study 223AS302 (NCTO1281189).
* Subjects of childbearing potential must practice effective contraception during the study and be willing and able to continue contraception for 1 month (females) or 3 months (males) after their last dose of study treatment.

Exclusion Criteria:

* Subject withdrew prematurely from Study CL211 (NCT00931944) or Study 223AS302 (NCTO1281189).
* Subject permanently discontinued study treatment in Study CL211 (NCT00931944) or Study 223AS302 (NCTO1281189) for any reason other than enrollment into this study.
* Subject from Study CL211 (NCT00931944) or Study 223AS302 (NCTO1281189) has a significant change in medical history (including laboratory tests or a clinically significant condition) that in the opinion of the Investigator would impair the subject's medical fitness for participation and preclude treatment.
* Female subject who is pregnant or breastfeeding.
* Subject is currently enrolled in any investigational drug study other than Study CL211 (NCT00931944) or Study 223AS302 (NCTO1281189).
* Subject is taking pramipexole, other dopamine agonists, any other agent with dopaminergic activity, or any other disallowed concomitant medication.
* Subject is unwilling or unable to comply with the requirements of the protocol including the presence of any condition (physical, mental, or social) that is likely to affect the subject's ability to comply with the protocol. At a minimum, subjects who are not able to travel to the study site must be willing to agree to remote blood draws for clinical laboratory evaluations and telephone visits to report Adverse Events, concomitant medications, and Amyotrophic Lateral Sclerosis Functional Rating Scale (revised) (ALSFRS-R) scores.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 616 (Actual)
Dates: Start 2012-06; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Bozik, MD, Study Chair — Knopp Biosciences
Locations (80):
- United States (42):
  - Barrow Neurological Institute - St. Joseph's Hospital, Phoenix, Arizona
  - University of California at San Francisco - Fresno, Fresno, California
  - University of California, Irvine, Orange, California
  - University of California, Davis, Sacramento, California
  - California Pacific Medical Center, San Francisco, California
  - Hospital for Special Care, New Britain, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - University of South Florida Medical Center, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Indiana University, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Charlestown, Massachusetts
  - St. Mary's Health Care, Grand Rapids, Michigan
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Neurology Associates, P.C., Lincoln, Nebraska
  - University of Nevada School of Medicine, Las Vegas, Nevada
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University, New York, New York
  - Research Foundation of the State University of New York, Syracuse, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Providence ALS Center, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - ALS Center at Penn, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Neurology, Dallas, Texas
  - Methodist Neurological Institute, Houston, Texas
  - University of Texas Health Sciences Center, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia Health System, Charlottesville, Virginia
  - University of Washington, Seattle, Washington
- Australia (4):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Royal Brisbane and Women's Hospital, Herston, Queensland
  - Calvary Health Care Bethlehem, Melbourne, Victoria
- Belgium (2):
  - AZ St-Lucas, Ghent
  - UZ Leuven, Leuven
- Canada (6):
  - Univ of Calgary / Foothills MC, Calgary, Alberta
  - CHUM - Hopital Notre Dame, Montreal, Quebec
  - Mcgill University, Montreal, Quebec
  - London Health Sciences Centre, London
  - Sunnybrook and Women's College and Health Sciences Centre, Toronto
  - University of British Columbia, Vancouver
- France (5):
  - CHRU de Lille - Hôpital Roger Salengro, Lille
  - Centre Hospitalier La Timone, Marseille
  - CHU Gui de Chauliac, Montpellier
  - CHU de Nice - Hôpital de l'Archet 1, Nice
  - Hôpital La Pitié Salpétrière, Paris
- Germany (5):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Bergmannsheil Gmbh, Bochum
  - Medizinische Hochschule Hannover (MHH), Hanover
  - Universitätsklinikum Jena, Jena
  - University of Ulm, RKU, Ulm
- Beaumont Hospital, Dublin, Ireland
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - UMC St. Radboud, Nijmegen
  - Universitair Medisch Centrum Utrecht, Utrecht
- Spain (4):
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - Hospital La Paz, Madrid
  - Hospital Carlos III, Madrid
- Sweden (2):
  - Sahlgrenska Universitetssjukhuset, Gothenburg
  - Karolinska Universitetssjukhuset, Solna, Stockholm
- United Kingdom (6):
  - Queen Elizabeth Hospital, Birmingham
  - Walton Centre for Neurology & Neurosurgery, Liverpool
  - Kings College Hospital NHS Foundation Trust, London
  - Newcastle University Hospital - Clinical Ageing Research Unit, Newcastle
  - John Radcliffe Hospital, Oxford
  - Sheffield Institute for Transnational Neuroscience, Sheffield

RESULTS

PARTICIPANT FLOW:
Groups:
- Dexpramipexole 300 mg/Day: Dexpramipexole: Oral tablet 150 mg given twice daily up to 36 months
Period: Overall Study
Arm/Group | Dexpramipexole 300 mg/Day
Started | 616
Completed | 0
Not Completed | 616
Not completed — Adverse Event | 20
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 20
Not completed — Investigator Decision | 1
Not completed — Death | 53
Not completed — STUDY TERMINATED EARLY BY SPONSOR | 521

BASELINE CHARACTERISTICS:
Population: This open-label extension study consisted of a Baseline Visit, a treatment period of up to 36 months, and a Safety Follow-Up Visit. Subjects who completed either Study CL211 or Study 223AS302 were eligible to participate in this study. If possible, the last visit of the lead-in study was used the Baseline. Otherwise, subjects were required to enroll within 14 days of their last visit in the lead-in study.
Groups:
- Dexpramipexole 150 mg BID: Dexpramipexole: Oral tablet 150 mg given twice daily up to 36 months
Arm/Group | Dexpramipexole 150 mg BID
Number analyzed (Participants) | 616
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One subject did not have age at Baseline reported.
  years
    number analyzed (Participants) | 615
    (all) | 56.5 (11.48)
Age, Customized [Count of Participants; unit: Participants]
  <50 years | 164
  between 50-65 years | 305
  >65 years | 146
  missing | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 206
  Male | 410
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 585
  More than one race | 0
  Unknown or Not Reported | 19
Region of Enrollment [Number; unit: participants]
  Canada | 39
  Netherlands | 26
  Sweden | 13
  Belgium | 21
  United States | 279
  Ireland | 14
  United Kingdom | 45
  Australia | 26
  France | 33
  Germany | 76
  Spain | 44
Weight (kg) [Mean (Standard Deviation); unit: kg] — Population: Weight was unable to be measured for many subjects due to ALS disease impairment (e.g., use of a mobility device).
  kg
    number analyzed (Participants) | 154
    (all) | 73.94 (16.528)
Height (cm) [Mean (Standard Deviation); unit: cm] | 173.1 (9.59)
Body mass index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — Population: Weight, and therefore BMI, was unable to be measured for many subjects due to ALS disease impairment (e.g., use of a mobility device).
  kg/m^2
    number analyzed (Participants) | 154
    (all) | 24.65 (5.058)

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Reported an Adverse Event
Description: The number of subjects who reported an adverse event during the study
Time Frame: Baseline through end of study (maximum 226 days: approximately 32.2 weeks)
Population: The safety population is defined as all subjects who received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dexpramipexole 150 mg BID
Number analyzed (Participants) | 616
Participants | 454

2. Primary Outcome: Number of Subjects Who Experienced a Serious Adverse Event
Description: The number of subjects enrolled who reported a serious adverse event during the study
Time Frame: Baseline through end of study (maximum 226 days: approximately 32.2 weeks)
Population: The safety population is defined as all subjects who received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dexpramipexole 150 mg BID
Number analyzed (Participants) | 616
Participants | 152

3. Primary Outcome: Number of Subjects Who Discontinued the Study Treatment Due to an Adverse Event
Description: The number of subjects enrolled who discontinued the study treatment due to an adverse event during the study
Time Frame: Baseline through end of study (maximum 226 days: approximately 32.2 weeks)
Population: The safety population is defined as all subjects who received at least 1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Dexpramipexole 150 mg BID
Number analyzed (Participants) | 616
Participants | 30

4. Primary Outcome: Number of Participants With Potentially Clinically Significant Vital Sign Results
Description: Number of Participants with Potentially Clinically Significant Vital Sign Abnormalities. Percentages based on number of patients with at least one non-missing post-baseline value in each treatment group. Patients are only counted once per criterion per laboratory test.
Time Frame: Baseline through end of study (maximum 226 days: approximately 32.2 weeks)
Population: The analysis population includes all subjects who received at least one dose of study drug and who had an evaluable post-baseline vital sign measurement during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexpramipexole 150 mg BID
Number analyzed (Participants) | 500
Participants
  Systolic BP >180 mmHg | 2
  Systolic BP Increase from Baseline >40 mmHg | 6
  Systolic BP <90 mmHg | 4
  Systolic BP Decrease from Baseline >30 mmHg | 10
  Diastolic BP >105 mmHg | 20
  Diastolic BP increase from Baseline >30 mmHg | 5
  Diastolic BP <50 mmHg | 2
  Diastolic BP Decrease from Baseline >20 mmHg | 21
  Pulse >120 bpm | 3
  Pulse Increase from Baseline >30 bpm | 16
  Pulse <50 bpm | 2
  Pulse Decrease from Baseline >20 bpm | 30
  Temperature >38.5 C and Increase from Baseline>=1°C: number analyzed (Participants) | 497
  Temperature >38.5 C and Increase from Baseline>=1°C | 1
  Weight >=7% Increase from Baseline: number analyzed (Participants) | 439
  Weight >=7% Increase from Baseline | 19
  Weight >=7% Decrease from Baseline: number analyzed (Participants) | 439
  Weight >=7% Decrease from Baseline | 37

5. Primary Outcome: Number of Participants With Potentially Clinically Significant Hematology Results
Description: Number of Participants with Potentially Clinically Significant Hematology Results. Percentages based on number of patients with at least one non-missing post-baseline value in each treatment group. Patients are only counted once per criterion per laboratory test.
Time Frame: Baseline through end of study (maximum 226 days: approximately 32.2 weeks)
Population: The analysis population includes all subjects who received at least one dose of study drug and who had an evaluable post-baseline hematology assessment during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexpramipexole 150 mg BID
Number analyzed (Participants) | 590
Participants
  White Blood Cell Count < 3.0 x10^9 cells/L | 18
  White Blood Cell Count >= 16 x10^9 cells/L | 6
  Total Absolute Neutrophil Count < 1.5 x10^9 cells/L | 14
  Total Absolute Neutrophil Count >= 13.5 x10^9 cells/L | 6
  Lymphocyte < 0.8 x10^9 cells/L | 65
  Lymphocyte > 12 x10^9 cells/L | 0
  Monocytes > 2.5 x10^9 cells/L | 0
  Eosinophils > 1.6 x10^9 cells/L | 0
  Basophils > 1.6 x10^9 cells/L | 0
  Hemoglobin - Females <= 95 g/L: number analyzed (Participants) | 194
  Hemoglobin - Females <= 95 g/L | 1
  Hemoglobin - Females >= 175 g/L: number analyzed (Participants) | 194
  Hemoglobin - Females >= 175 g/L | 0
  Hemoglobin - Males <= 115 g/L: number analyzed (Participants) | 396
  Hemoglobin - Males <= 115 g/L | 13
  Hemoglobin - Males >= 190 g/L: number analyzed (Participants) | 396
  Hemoglobin - Males >= 190 g/L | 1
  Hematocrit - Females <= 32%: number analyzed (Participants) | 194
  Hematocrit - Females <= 32% | 8
  Hematocrit - Females >= 54%: number analyzed (Participants) | 194
  Hematocrit - Females >= 54% | 0
  Hematocrit - Males <= 37%: number analyzed (Participants) | 396
  Hematocrit - Males <= 37% | 47
  Hematocrit - Males >= 60%: number analyzed (Participants) | 396
  Hematocrit - Males >= 60% | 1
  Red Blood Cell Count <= 3.5 x10^12 cells/L | 15
  Red Blood Cell Count >= 6.4 x10^12 cells/L | 3
  Platelet Count <= 75 x10^9 cells/L | 0
  Platelet Count >= 700 x10^9 cells/L | 3

6. Primary Outcome: Number of Participants With Potentially Clinically Significant Blood Chemistry Results
Description: Number of Participants with Potentially Clinically Significant Blood Chemistry Results. Percentages based on number of patients with at least one non-missing post-baseline value in each treatment group. Patients are only counted once per criterion per laboratory test.
Time Frame: Baseline through end of study (maximum 226 days: approximately 32.2 weeks)
Population: The analysis population includes all subjects who received at least one dose of study drug and who had an evaluable post-baseline blood chemistry assessment during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexpramipexole 150 mg BID
Number analyzed (Participants) | 589
Participants
  Sodium <= 126 mmol/L: number analyzed (Participants) | 588
  Sodium <= 126 mmol/L | 5
  Sodium >= 156 mmol/L: number analyzed (Participants) | 588
  Sodium >= 156 mmol/L | 0
  Potassium <= 3 mmol/L: number analyzed (Participants) | 587
  Potassium <= 3 mmol/L | 1
  Potassium >= 6 mmol/L: number analyzed (Participants) | 587
  Potassium >= 6 mmol/L | 4
  Chloride <= 90 mmol/L: number analyzed (Participants) | 588
  Chloride <= 90 mmol/L | 9
  Chloride >= 118 mmol/L: number analyzed (Participants) | 588
  Chloride >= 118 mmol/L | 0
  Bicarbonate <= 16 mmol/L: number analyzed (Participants) | 588
  Bicarbonate <= 16 mmol/L | 7
  Bicarbonate >= 35 mmol/L: number analyzed (Participants) | 588
  Bicarbonate >= 35 mmol/L | 6
  Calcium <= 2 mmol/L | 7
  Calcium >= 3 mmol/L | 0
  Magnesium <= 0.5 mmol/L: number analyzed (Participants) | 588
  Magnesium <= 0.5 mmol/L | 0
  Magnesium >= 1.2 mmol/L: number analyzed (Participants) | 588
  Magnesium >= 1.2 mmol/L | 0
  Phosphorus <= 0.6 mmol/L | 0
  Phosphorus >= 1.7 mmol/L | 9
  Aspartate Aminotransferase - SGOT >= 3 x ULN U/L: number analyzed (Participants) | 587
  Aspartate Aminotransferase - SGOT >= 3 x ULN U/L | 4
  Alanine Aminotransferase - SGPT >= 3 x ULN U/L: number analyzed (Participants) | 588
  Alanine Aminotransferase - SGPT >= 3 x ULN U/L | 12
  Alkaline Phosphatase >= 1.5 x ULN U/L | 4
  Creatinine - Females >= 176.8 umol/L: number analyzed (Participants) | 193
  Creatinine - Females >= 176.8 umol/L | 1
  Creatinine - Males >= 176.8 umol/L: number analyzed (Participants) | 396
  Creatinine - Males >= 176.8 umol/L | 0
  Blood Urea Nitrogen >= 10.7 mmol/L | 23
  Total Bilirubin >= 1.5 x ULN umol/L | 8
  Total Protein <= 45 g/L | 1
  Total Protein >= 100 g/L | 0
  Albumin <= 25 g/L | 3
  Uric Acid - Females >= 506 umol/L: number analyzed (Participants) | 193
  Uric Acid - Females >= 506 umol/L | 1
  Uric Acid - Males >= 625 umol/L: number analyzed (Participants) | 396
  Uric Acid - Males >= 625 umol/L | 4
  Glucose <= 2.2 mmol/L | 0
  Glucose >= 9.7 mmol/L | 43

7. Primary Outcome: Number of Participants With Potentially Clinically Significant ECG Results
Description: Number of Participants with Potentially Clinically Significant ECG Results. Percentages based on number of patients with at least one non-missing post-baseline value in each treatment group. Patients are only counted once per criterion per laboratory test.
Time Frame: Baseline through end of study (maximum 226 days: approximately 32.2 weeks)
Population: The analysis population includes all subjects who received at least one dose of study drug and who had an evaluable post-baseline ECG assessment during the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dexpramipexole 150 mg BID
Number analyzed (Participants) | 460
Participants
  QTcF > 450 ms | 2
  QTcF > 480 ms | 0
  QTcF > 500 ms | 0
  QTcF Change from Baseline > 30 ms: number analyzed (Participants) | 457
  QTcF Change from Baseline > 30 ms | 34
  QTcF Change from Baseline > 60 ms: number analyzed (Participants) | 457
  QTcF Change from Baseline > 60 ms | 3
  QT > 450 ms | 0
  QT > 480 ms | 0
  QT > 500 ms | 0
  QT Change from Baseline > 30 ms: number analyzed (Participants) | 457
  QT Change from Baseline > 30 ms | 59
  QT Change from Baseline > 60 ms: number analyzed (Participants) | 457
  QT Change from Baseline > 60 ms | 2
  QTcB > 480 ms | 9
  QTcB > 450 ms | 2
  QTcB > 500 ms | 0
  QTcB Change from Baseline > 30 ms: number analyzed (Participants) | 457
  QTcB Change from Baseline > 30 ms | 69
  QTcB Change from Baseline > 60 ms: number analyzed (Participants) | 457
  QTcB Change from Baseline > 60 ms | 6
  PR > 220 ms and Percent Increase from Baseline >25%: number analyzed (Participants) | 455
  PR > 220 ms and Percent Increase from Baseline >25% | 0
  QRS > 110 ms and Percent Increase from Baseline >25%: number analyzed (Participants) | 457
  QRS > 110 ms and Percent Increase from Baseline >25% | 1

8. Secondary Outcome: Slope of ALSFRS-R (ALS Functional Rating Scale With Respiratory Component) From Baseline to End of Study
Description: The ALSFRS-R (ALS functional rating scale with respiratory component) is a validated scale which measures 4 functional domains, comprising respiratory function, bulbar function, gross motor skills, and fine motor skills. There are a total of 12 questions, each scored from 0 to 4 for a total possible score between 0 to 48, with higher scores representing better function. Slope is calculated using a linear mixed effects model with x-axis time in months and y-axis ALSFRS-R score. Units for slope are change per month in units on the ALSFRS-R scale.
Time Frame: Up to maximum 226 days: approximately 32.2 weeks
Population: Randomized subjects who had at least 1 post-baseline clinical evaluation
Measure: Least Squares Mean (Standard Error); unit: Change per month in ALSFRS-R
Groups:
- Dexpramipexole 150 mg BID: Dexpramipexole: Oral tablet 150 mg given twice daily up to 7 months
Arm/Group | Dexpramipexole 150 mg BID
Number analyzed (Participants) | 607
Change per month in ALSFRS-R | -0.7355 (0.04448)

9. Secondary Outcome: Slope of Sniff Nasal Inspiratory Pressure (SNIP) From Baseline to End of Study
Description: SNIP is a test of inspiratory force (sternocleidomastoid and diaphragm) measured via a nasal cannula and is used to assess respiratory muscle weakness and to monitor changes in respiratory muscle strength over time. During the SNIP maneuver, the patient is asked to perform a strong, sharp, maximal sniff, whereby nasal pressure is measured via nasal cannula. The maximum recorded value after several attempts, with rest in between attempts, was use in the analysis.
Time Frame: Up to maximum 226 days: approximately 32.2 weeks
Population: Randomized subjects who had at least 1 post-baseline clinical evaluation
Measure: Least Squares Mean (Standard Error); unit: Change per month in SNIP (in cm H20)
Arm/Group | Dexpramipexole 150 mg BID
Number analyzed (Participants) | 610
Change per month in SNIP (in cm H20) | -0.1895 (0.09933)

10. Secondary Outcome: Death up to 6 Months
Description: Kaplan-Meier estimate of percentage of subjects who died up to 6 months
Time Frame: 6 Months
Population: Subjects who were randomized, received at least 1 dose of study treatment, had at least 1 available post-dosing efficacy evaluation (ALSFRS-R) or died during the study period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dexpramipexole 150 mg BID
Number analyzed (Participants) | 615
percentage of participants | 13.95 [10.83 to 17.07]

11. Secondary Outcome: Percentage of Participants With Death or Death Equivalent up to 6 Months
Description: Kaplan-Meier estimate of percentage of subjects who died or had a death equivalent event (tracheostomy or permanent assisted ventilation [PAV], defined as use of noninvasive ventilation [NIV] for ≥22 hours per day for ≥10 days) up to 6 months
Time Frame: 6 months
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dexpramipexole 150 mg BID
Number analyzed (Participants) | 615
percentage of participants | 16.35 [13.00 to 19.70]

ADVERSE EVENTS:
Time Frame: Adverse events were collected between the time of the first dose of study treatment and the last study visit for each enrolled subject. In this study, the maximum subject duration was a maximum 226 days: approximately 32.2 weeks.
Arm/Group | Dexpramipexole 300 mg/Day
All-Cause Mortality (participants affected / at risk) | 73/616
Serious Adverse Events (participants affected / at risk) | 152/616
Other Adverse Events (participants affected / at risk) | 215/616
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dexpramipexole 300 mg/Day (N=616)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1
LEUKOPENIA (Blood and lymphatic system disorders) | 1
NEUTROPENIA (Blood and lymphatic system disorders) | 2
CARDIAC ARREST (Cardiac disorders) | 2
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 1
STRESS CARDIOMYOPATHY (Cardiac disorders) | 1
VENTRICULAR FIBRILLATION (Cardiac disorders) | 1
COLITIS (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
DYSPHAGIA (Gastrointestinal disorders) | 16
FAECALOMA (Gastrointestinal disorders) | 1
GASTROINTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1
DEATH (General disorders) | 1
EUTHANASIA (General disorders) | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1
HAEMORRHOIDS (General disorders) | 1
PYREXIA (General disorders) | 1
CHOLECYSTITIS (Hepatobiliary disorders) | 1
BRONCHITIS (Infections and infestations) | 1
CATHETER SITE INFECTION (Infections and infestations) | 1
CLOSTRIDIUM DIFFICILE COLITIS (Infections and infestations) | 1
ENTEROCOCCAL INFECTION (Infections and infestations) | 1
ENTEROCOCCAL SEPSIS (Infections and infestations) | 1
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1
GASTROENTERITIS (Infections and infestations) | 1
HERPES ZOSTER OTICUS (Infections and infestations) | 1
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1
ORAL INFECTION (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 15
PNEUMONIA PNEUMOCOCCAL (Infections and infestations) | 1
PSEUDOMONAL BACTERAEMIA (Infections and infestations) | 1
RESPIRATORY TRACT INFECTION (Infections and infestations) | 2
UROSEPSIS (Infections and infestations) | 2
CAPNOTHORAX (Injury, poisoning and procedural complications) | 1
CERVICAL VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 1
FALL (Injury, poisoning and procedural complications) | 3
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1
HIP FRACTURE (Injury, poisoning and procedural complications) | 1
BLOOD GLUCOSE INCREASED (Investigations) | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 1
SLEEP STUDY (Investigations) | 2
WEIGHT DECREASED (Investigations) | 2
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 2
BRONCHIAL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
AMYOTROPHIC LATERAL SCLEROSIS (Nervous system disorders) | 16
ANXIETY (Psychiatric disorders) | 2
CONFUSIONAL STATE (Psychiatric disorders) | 1
HALLUCINATION (Psychiatric disorders) | 1
CALCULUS URETERIC (Renal and urinary disorders) | 1
HYDRONEPHROSIS (Renal and urinary disorders) | 1
URINARY RETENTION (Renal and urinary disorders) | 1
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 2
ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1
CHRONIC RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 4
FOREIGN BODY ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 1
HYPOVENTILATION (Respiratory, thoracic and mediastinal disorders) | 1
LARYNGOSPASM (Respiratory, thoracic and mediastinal disorders) | 1
NASAL SEPTUM DEVIATION (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONIA ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 5
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 1
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 3
RESPIRATORY ARREST (Respiratory, thoracic and mediastinal disorders) | 2
RESPIRATORY DISORDER (Respiratory, thoracic and mediastinal disorders) | 1
RESPIRATORY DISTRESS (Respiratory, thoracic and mediastinal disorders) | 2
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 50
RESPIRATORY MUSCLE WEAKNESS (Respiratory, thoracic and mediastinal disorders) | 1
ANGIOEDEMA (Skin and subcutaneous tissue disorders) | 1
RASH GENERALISED (Skin and subcutaneous tissue disorders) | 1
RESPITE CARE (Social circumstances) | 1
GASTROSTOMY TUBE INSERTION (Surgical and medical procedures) | 1
INTESTINAL RESECTION (Surgical and medical procedures) | 1
MECHANICAL VENTILATION (Surgical and medical procedures) | 1
TRACHEOSTOMY (Surgical and medical procedures) | 2
DEEP VEIN THROMBOSIS (Vascular disorders) | 2
SHOCK (Vascular disorders) | 1
THROMBOSIS (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dexpramipexole 300 mg/Day (N=616)
URINARY TRACT INFECTION (Infections and infestations) | 31
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 52
CONSTIPATION (Gastrointestinal disorders) | 49
NAUSEA (Gastrointestinal disorders) | 33
OEDEMA PERIPHERAL (General disorders) | 31
FALL (Injury, poisoning and procedural complications) | 68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must be consulted